CLINICAL TRIAL: NCT03039088
Title: PREDICT-SpA - French Epidemiological Study of the Evaluation of the Impact of Fibromyalgia in the TNF Alpha Treatment Effect in Axial Spondyloarthritis in Both Anti-TNF naïve and - Experienced Patients
Acronym: PREDICT_SpA
Status: Completed | Type: Observational
Sponsor: Association de Recherche Clinique en Rhumatologie (Other)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-A01288-39
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-01

CONDITIONS: Axial Spondyloarthritis; Fibromyalgia
MeSH Terms: conditions — Axial Spondyloarthritis; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia patients
  Interventions: Other: Follow-up after 12 weeks after TNF alpha blockers initiation
- Not fibromyalgia patients
  Interventions: Other: Follow-up after 12 weeks after TNF alpha blockers initiation

INTERVENTIONS:
Other: Follow-up after 12 weeks after TNF alpha blockers initiation

SUMMARY:
This is a prospective observational national (France) study with 2 visits 3 months apart (baseline and 12 weeks after TNF alpha blockers initiation). The objective of recruitment is 500 SpA patients (diagnosis according to their treating rheumatologist) initiating a TNF alpha blocker.

The main objective of the study is to evaluate the impact of a concomitant fibromyalgia on the anti-TNF treatment effect in axial Spondyloarthritis in both anti-TNF naïve and pre-exposed patients.

DETAILED DESCRIPTION:
Background: Diagnosis of SpA in the absence of objective signs of inflammation or structural damage can be challenging, and especially difficult to differentiate from Fibromyalgia. Furthermore, such patients can easily be classified as active and refractory to NSAIDs, and inappropriately receive TNF alpha blockers.

Objective: Primary objective: To evaluate the impact of fibromyalgia in the TNF alpha treatment effect in axial Spondyloarthritis in both anti-TNF naïve and - experienced patients.

Methods: Design: Prospective observational national (France) study with 2 visits 3 months apart (baseline and 12 weeks after TNF alpha blockers initiation). Patients: 500 SpA patients (diagnosis according to their treating rheumatologist) initiating a TNF alpha blocker. Data collection: items permitting the calculation of the ASAS criteria, the FIRST questionnaire (Fibromyalgia Rapid Screen Test), patients and disease characteristics, disease activity and severity items, and the domain leading the doctor's decision for initiating the TNF alpha blocker (CRP/Imaging/Symptoms) will be collected at baseline. Effectiveness measures (e.g. BASDAI and patient's global) and the doctor's decision to continue/discontinue the TNF alpha blocker will be collected during the second visit. Statistical analysis: for the main objective, evaluation of the predictive factors of a TNF alpha response in real life, and the impact of Fibromyalgia in such response (e.g. logistic regression to estimate BASDAI reduction of 50%). For the secondary objectives: evaluation of the relative attributable risks of the doctor's domains leading the TNF alpha blocker initiation (Imaging/CRP/Symptoms) in order to explain the anti-TNF therapy response; evaluation of the concordance existing between the current recommendations and the daily practice.

Expected results: A positive finding might results into a change in the way of managing patients (e.g. carefully checking for the co-existence of fibromyalgia before confirming a spondyloarthritis diagnosis, an active disease and also before initiating a specific therapy such as biologics.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years old and suffering from SpA based on the opinion of the treating rheumatologist
* Patients in whom the decision of initiating of switching an anti-TNF because of an axial involvement of SpA has been made by the treating rheumatologist. In case of previous exposure to antiTNF a washout period of at least 4 weeks be asked.

Exclusion Criteria:

* Patients unable to understand the questionnaire
* Patients not giving their informed written consent
* Patients with absolute contraindications to anti-TNF as per label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from SpA based on the opinion of the treating rheumatologist initiating a TNF alpha blocker.
Sampling Method: Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamitouche F, Lopez-Medina C, Gossec L, Perrot S, Dougados M, Molto A. Evaluation of the agreement between the ACR 1990 fibromyalgia tender points and an enthesitis score in patients with axial spondyloarthritis. Rheumatology (Oxford). 2023 Aug 1;62(8):2757-2764. doi: 10.1093/rheumatology/keac683. PMID 36573318

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibromyalgia Patients: 202 (38.4%) according to the FiRST questionnaire.
- Not Fibromyalgia Patients: 324 (61.6%) according to the FiRST questionnaire
Period: Overall Study
Arm/Group | Fibromyalgia Patients | Not Fibromyalgia Patients
Started | 192 | 316
Completed | 192 | 316
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fibromyalgia Patients; Not Fibromyalgia Patients: According to the FiRST Questionnaire
  Follow-up after 12 weeks after TNF alpha blockers initiation
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia Patients | Not Fibromyalgia Patients | Total
Number analyzed (Participants) | 202 | 324 | 526
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 202 | 324 | 526
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.7) | 41.1 (12.1) | 41.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 134 | 245
  Male | 91 | 190 | 281

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Presence of Fibromyalgia (Defined by a FIRST Questionnaire >= 5/6) as a Predisposing Factor for Lower Treatment Response Rates to TNF Alpha Blockers
Description: The difference in BASDAI50 response at week 12 between the patients with and those without fibromyalgia.
Time Frame: At 12 weeks after TNF alpha blockers initiation
Measure: Number; unit: participants
Groups:
- Fibromyalgia Patients: 192 (37.8%) according to the FiRST questionnaire.
Arm/Group | Fibromyalgia Patients | Not Fibromyalgia Patients
Number analyzed (Participants) | 192 | 316
participants | 87 | 171

2. Secondary Outcome: The Relative Attributable Risks of the Doctor's Reported Outcomes Versus the Patients Reported Outcomes in the Decision to Initiate/Switch Anti-TNF Therapy
Time Frame: At 12 weeks after TNF alpha blockers initiation
Reporting Status: Not Posted

3. Secondary Outcome: Pourcentage of Patients With Fibromyalgia (as Co-morbidity or as Single Disease)
Time Frame: At 12 weeks after TNF alpha blockers initiation
Reporting Status: Not Posted

4. Secondary Outcome: Evaluation of the Concordance Existing Between the Current Recommendations for the Initiation of Anti-TNF in Non-radiographic Axial SpA and the Daily Practice as Represented by This Study.
Time Frame: At baseline and at 12 weeks after TNF alpha blockers initiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Fibromyalgia Patients | Not Fibromyalgia Patients
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/324
Other Adverse Events (participants affected / at risk) | 0/202 | 0/324

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No